CLINICAL TRIAL: NCT00901615
Title: A Phase IB Study of Escalating Doses of REVLIMID in Association With R-CHOP (R2-CHOP) in the Treatment of B-cell Lymphoma
Brief Title: Lenalidomide and R-CHOP in B-cell Lymphoma
Acronym: R2CHOP-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2CHOP-1
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma
Keywords: lymphoma; lenalidomide; gela
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide and R-CHOP (Experimental): Escalating Lenalidomide dose from 2.5 to 25 mg Lenalidomide and R-CHOP
  Interventions: Drug: Lenalidomide and R-CHOP

INTERVENTIONS:
Drug: Lenalidomide and R-CHOP — Lenalidomide dose administered orally during 14 days in combination with 6 courses of fixed doses of R-CHOP 21.
  Other Names: REVLIMID

SUMMARY:
The purpose of the study is to determine the recommended dose (RD) of lenalidomide (Revlimid) when administered in association with R-CHOP (rituximab (R), cyclophosphamide, doxorubicin, vincristine and prednisone).

DETAILED DESCRIPTION:
The study is a dose escalation study of lenalidomide (Revlimid) administered orally during 14 days in combination with fixed doses of rituximab (R), cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered every 3 weeks (R-CHOP 21) in patients with B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of the following B-cell Lymphoma, CD 20 positive:

  * Mantle cell, Marginal zone, follicular
  * Histological transformation from low grade to high grade
  * Diffuse large B cell
* Aged from 18 to 70 years
* WHO performance status 0, 1 or 2
* Signed inform consent
* Life expectancy of ≥ 90 days (3 months).
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL not more than 3 days from the start of study drug and must either commit to continued abstinence from heterosexual intercourse or begin one acceptable method of birth control, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to monthly pregnancy testing and must be counseled at a minimum of every 4 weeks about pregnancy precautions and risks of fetal exposure.
* Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential. Men must also be counseled at a minimum of every 4 weeks about pregnancy precautions and risks of fetal exposure.

  * † A female patient is considered to have childbearing potential unless she meets at least one of the following criteria 1) Age > 50 years and naturally amenorrhoeic for > 1 year (amenorrhoea following cancer therapy does not rule out childbearing potential); or 2) Premature ovarian failure confirmed by a specialist gynaecologist or 3) Previous bilateral salpingo-oophorectomy, or hysterectomy, or 4) XY genotype, turner syndrome, uterine agenesis.

Exclusion Criteria:

* Previous treatment with immunotherapy or chemotherapy except:

  * Chlorambucil or Cyclophosphamide per os alone during less than 6 months, if stopped more than one year before inclusion
  * Rituximab alone during less than three months, if stopped more than one year before inclusion
* Previous radiotherapy except if localized to one lymph node area
* Other type of lymphomas: Burkitt, T cell, lymphocytic, CD 20 negative
* Central nervous system or meningeal involvement
* Contraindication to any drug contained in the chemotherapy regimen
* HIV disease, active hepatitis B or C
* Any serious active disease or co-morbid medical condition (according to investigator's decision)
* Any of the following laboratory abnormalities :

  * Absolute neutrophil count (ANC) < 1,500 cells/mm3 (1.5 x 109/L).
  * Platelet count < 100,000/mm3 (100 x 109/L).
  * Serum SGOT/AST or SGPT/ALT 5.0 x upper limit of normal (ULN).
  * Serum total bilirubin > 2.0 mg/dL (34 µmol/L), except in case of hemolytic anemia.
* Calculated creatinine clearance (Cockcroft-Gault formula) of < 50 mL /min
* Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 3 years
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females.
* Prior ≥ Grade 3 allergic reaction/hypersensitivity to thalidomide.
* Prior ≥ Grade 3 rash or any desquamating (blistering) rash while taking thalidomide.
* Subjects with ≥ Grade 2 neuropathy.
* Prior use of lenalidomide.
* Use of any standard or experimental anti-cancer drug therapy within 28 days of the initiation (Day 1) of study drug therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-01-06 (Actual); Primary Completion 2010-11-19 (Actual); Study Completion 2015-11-23 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | 42 days

SECONDARY OUTCOMES:
Complete response rate and Overall response rate at the end of treatment | 3 months after the end of treatment
Complete and Overall response rates after induction | at the end of third cycle of treatment (between Day 56 and Day 63)
Progression-Free Survival and Overall survival | 7 years
Duration of response | 7 years
Collection of adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hervé TILLY, Prof, Principal Investigator — Lymphoma Study Association
Locations (5):
- France (5):
  - CHU de Dijon, Dijon
  - CHRU Lille, Lille
  - CHU Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - CHU Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- See also: GELA — http://www.gela.org